CLINICAL TRIAL: NCT06401811
Title: Reliability, Validity, and Responsiveness of the Turkish Version of Eating Assessment Tool-10 for Patients With Primer Sjögren's Syndrome
Status: Recruiting | Type: Observational
Sponsor: Kahramanmaras Sutcu Imam University (Other)
Responsible Party: Principal Investigator, Nazli Elif Nacar, Lecturer, Kahramanmaras Sutcu Imam University
Other Study IDs: KSU.
Record Dates: First submitted 2024-05-02; First posted 2024-05-07 (Actual); Last update posted 2024-06-25 (Actual); Status verified 2024-06

CONDITIONS: Sjogren's Syndrome
Keywords: Primer Sjogren's Syndrome; swallowing disorder
MeSH Terms: conditions — Sjogren's Syndrome; Deglutition Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Evaluations will be made by researchers following the guidance of individuals with primary Sjögren's Syndrome who receive diagnosis, routine medical care, and treatment management.

In addition, for the reliability of the Turkish Eating Assessment Tool-10, the Turkish Eating Assessment Tool-10 will be repeated on patients at least one-fifth of the number of individuals included, after one week.

For the sensitivity of the scale, an exercise that is routinely applied in the Rheumatological Rehabilitation Unit of Hacettepe University Faculty of Physical Therapy and Rehabilitation will be invited and after 3 months, the same evaluations as applied in the first measurement will be made again on individuals at least one-fifth of the number of individuals included.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with Primary Sjögren's Syndrome
* 18 years or older

Exclusion Criteria:

* Patients with Secondary Sjögren's Syndrome,
* Patients who are diagnosed with other uncontrolled/clinically important diseases (chronic obstructive pulmonary disease, congestive heart failure, endocrine system diseases, neurological, psychological diseases, etc.),
* Individuals who do not agree to participate in the study and do not give written consent will be excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with primer Sjogren's Syndrome diagnosed by a rheumatologist.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-06-04 (Actual); Primary Completion 2024-08-30 (Estimated); Study Completion 2024-11-30 (Estimated)

PRIMARY OUTCOMES:
Turkish Eating Assessment Tool | Baseline-first week-third month
  Turkish Eating Assessment Tool-10 is a survey consisting of 10 questions with a Likert scale between 0 and 4 (0 = no problem, 4 = severe problem). The total score is calculated out of 40 points by finding the sum of the answers given by individuals to each question. A score of 3 or more in the survey is considered abnormal. A score of 16 or above is considered a suspicion of aspiration. Turkish validity and reliability were tested by authors in 2016.

SECONDARY OUTCOMES:
Yale Swallow Protocol | Baseline-third month
  Yale Swallow Protocol is a reliable screening test performed under expert supervision to determine the risk of aspiration at an early stage. The protocol has three main components. These are exclusion criteria, a short cognitive test, and oral mechanism, and drinking 3 oz (90 cc) water directly from the glass or with a straw. Risk factors are examined in the 1st and 2nd stages to determine the patients to whom the test can be applied. Patients who complete step 1 and are not contraindicated for testing proceed to the short cognitive testing phase. Patients who pass the short cognitive test and oral mechanism stages can proceed to the third stage, which is drinking 90 cc of water. The 90 cc water swallow challenge protocol is a simple assessment that can be used by many qualified healthcare professionals to identify aspiration risk because it is easy to perform, highly reliable, cost-effective, and clinically validated.Patients showing these findings are recorded as 'failing' the test.

OTHER OUTCOMES:
Test of Mastication and Swallowing Solids | Baseline-third month
  In our study, the Test of Mastication and Swallowing Solids (TOMASS) will be used. The test evaluates how many bites the individual takes to eat a biscuit while sitting upright, how many chewing cycles he makes, how many times he swallows it, and how long the total time is from biting to swallowing. Video recording will be taken during the test. The number of bites, number of chewing cycles, number of swallows and total time will be calculated on the video. Individuals will be asked to eat the biscuit normally while sitting on a chair in an upright position with the throat visible. Meanwhile, video recording will be taken from the individuals' front view, showing their mouth and neck. The evaluation of the test will then be made by the evaluator. Videos will be stored in folders on an encrypted computer and only the work team will have access.
Dysphagia limit | Baseline-third month
  While evaluating dysphagia, individuals are given 5, 10, 15, 20, 25, 30, 35, 40 and 45 mL volumes of liquid, respectively, with a graduated syringe and are asked to swallow the liquid. The maximum amount of fluid that the thyroid cartilage can swallow during a single movement is determined. The normal dysphagia limit in healthy individuals is more than 20 mL. If a person can swallow 20 mL normally, the dysphagia limit is normal.

CONTACTS AND LOCATIONS:
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)